CLINICAL TRIAL: NCT06954779
Title: Arginine Plaque Metabolism Pilot Clinical Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2023-SAL-05-EG
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Plaque, Dental
Keywords: saliva
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test 1 toothpaste (Active Comparator): fluoride toothpaste
  Interventions: Drug: Colgate Cavity Protection
- Test 2 toothpaste (Experimental): non fluoride toothpaste
  Interventions: Drug: TOM's Superior Sensitivity Relief Toothpaste

INTERVENTIONS:
Drug: Colgate Cavity Protection — 1000ppm fluoride
  Arms: Test 1 toothpaste
Drug: TOM's Superior Sensitivity Relief Toothpaste — fluoride free
  Arms: Test 2 toothpaste

SUMMARY:
Proof of concept clinical study to measure plaque metabolism and the prebiotic efficacy of arginine-containing toothpaste.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects aged 18-70 years, inclusive.
* Availability for the nine-week duration of the clinical research study.
* Good general health based on the opinion of the study investigator
* Good general health

Exclusion Criteria:

* Moderate and/or advanced periodontal disease, rampant caries, or any condition that the dental examiner considers exclusionary from the study.
* Five or more carious lesions requiring immediate care.
* Concurrent participation in any other oral care clinical study or test panel.
* Self-reported pregnant or lactating women.
* Dental prophylaxis received in the past four weeks prior to baseline examinations
* History of tobacco use-smoking, vaping and chewing tobacco
* Presence of orthodontic bands, presence of partial removable dentures
* Tumor(s) of the soft or hard tissues of the oral cavity
* Use of antibiotics or stain inducing medications any time during the two month prior to entry into the study
* Use of oral care products containing antimicrobials (Zn, Sn, CPC, triclosan, alcohol containing mouthwash, etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Plaque collection | baseline, week 3, week 4, week 6, week 7, week 8, week 9
  Fasting plaque will be collected before and after a sucrose rinse for lactic acid analysis and ammonia production.The plaque pH of collected samples will also be measured to provide trend data.

SECONDARY OUTCOMES:
Saliva collection | week 5 and week 9
  Differences in the arginine concentration in saliva pre- and post-brushing with treatment. Differences in microbiome composition and activity

CONTACTS AND LOCATIONS:
Locations (1):
- Volpe Clinical Center, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No